CLINICAL TRIAL: NCT01820377
Title: Northern Lights Physical Activity Program for Management of Type 2 Diabetes Early in Life: Aboriginal Youth Mentorship Program
Brief Title: The Aboriginal Youth Mentorship Program
Acronym: AYMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Institute of Child Health (Industry); The Lawson Foundation (Other)
Responsible Party: Principal Investigator, Jon McGavock, Associate Professor, University of Manitoba
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: H2008:060
Record Dates: First submitted 2013-03-21; First posted 2013-03-28 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Peer-mentoring; Obesity; Type 2 Diabetes; Physical Activity; After-school program
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aboriginal Youth Mentorship Program (Experimental): High school students volunteer as mentors, and develop an after-school program that they then deliver to children in grade 4. The mentors meet twice a week. The first day, they develop an activity plan and decide roles and responsibilities to ensure successful delivery of each activity. The second day, they deliver the program to the grade 4 students, which incorporates a healthy snack, 45-minutes of physical activity, and educational games/activities. Grade 4s act as the intervention group.
  Interventions: Behavioral: Aboriginal Youth Mentorship Program
- Control Group (No Intervention): This group acts as a control, and are not apart of the Aboriginal Youth Mentorship Program

INTERVENTIONS:
Behavioral: Aboriginal Youth Mentorship Program — High school students volunteer as mentors, and develop an after-school program that they then deliver to children in grade 4. The mentors meet twice a week. The first day, they develop an activity plan and decide roles and responsibilities to ensure successful delivery of each activity. The second day, they deliver the program to the grade 4s, which incorporates a healthy snack, 45-minutes of physical activity, and educational games/activities. Grade 4s are our intervention group
  Other Names: AYMP
  Arms: Aboriginal Youth Mentorship Program

SUMMARY:
Building on the successes of a communal, relationship based approach to Aboriginal youth mentoring in an after school physical activity program (AYMP), the investigators are evaluating a peer-led approach for diabetes prevention.

DETAILED DESCRIPTION:
Building on the successes of a communal, relationship based approach to Aboriginal youth mentoring in an after school physical activity program (AYMP), the investigators are evaluating a peer-led approach for diabetes prevention. High school students volunteer as mentors, and develop an after-school program that they then deliver to children in grade 4. The mentors meet twice a week. The first day, they develop an activity plan and decide roles and responsibilities to ensure successful delivery of each activity. The second day, they deliver the program to the grade 4s, which incorporates a healthy snack, 45-minutes of physical activity, and educational games/activities. Our primary goal is to determine the health benefits of AYMP; guided by our youth mentors and community advisors, the investigators will also develop a number of research questions that will help us to better understand the social, emotional, physical and spiritual outcomes of the peer-led mentor program. To answer these questions, the investigators will train community members in both qualitative and quantitative methods. The quantitative outcomes of this study include physical activity, waist circumference, obesity rates, and self-esteem. Qualitative methods may include photovoice and focus group interviews. All of these will be used to assess the social determinants of health and contextual features of the program.

ELIGIBILITY:
Inclusion Criteria:

* Grade 4 students. We chose to intervene with youth in grade 4 for four primary reasons: (1) the large majority of youth in grade 4 are in tanner stage 1 and will not experience puberty-related weight gain during the school year; (2) previous experience by our group revealed that attendance throughout the school year is higher in students in grade 4 relative to students in grade 5 or 6; (3) students in grade 4 are old enough to perform low organized games included in the intervention; and (4) retention rates in the intervention are greater than students in grades 5 and 6.

Exclusion Criteria:

* While all students will be invited to participate in the intervention, for measurement purposes, we will exclude data from those students who may not respond to the intervention or would be unable to participate in the physical activity aspects of the component. This includes children with: (1) musculoskeletal injuries that limit physical activities; (2) treatment for chronic conditions that would elicit weight gain or limit participation in physical activity (insulin, corticosteroids, blood pressure medications); (3) poor attendance (<60% of school days) in the first semester; (4) children whose parents are unwilling to provide consent. Note: the intervention will be offered to youth with chronic conditions, however their data will not be included in the final analysis, due to confounding effects of medications.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 246 (Actual)
Dates: Start 2010-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Waist Circumference | 5 months
  The primary outcome will be waist circumference measured at the level of the iliac crest. Waist circumference is a clinically relevant outcome as it is a robust predictor of Type 2 Diabetes in youth and other cardiometabolic outcomes in youth.

SECONDARY OUTCOMES:
Daily Physical Activity | 5 months
  The secondary outcomes include daily physical activity measured using a pedometer
Rates of overweight/obesity between groups | 5 months
  Rates of overweight and obesity between the groups will be measured before and after the intervention
Self-Efficacy in Peer Interactions | 5 months
  This scale is designed to measure youths' perceptions of their ability to be successful in social interactions. This includes their ability to be persuasive towards peers in positive ways. The questionnaire contains two subscales that measure social self-efficacy in conflict and non-conflict situations. The subscales can be used separately or combined into a total score.
Civic Responsibility Survey | 5 months
  This scale measures youths' community awareness, knowledge, and investment in helping to improve their community.
Teacher-on-Pupil Strengths and Difficulties Questionnaire | 5 months
  The Teacher on Pupil Questionnaire for the Child Cohort recorded specific information about the Study child, such as temperament, academic performance and school preparedness.
Parent Lifestyle Behaviours Questionnaire | 5 months
  Questions about Socioeconomic status, as well as daily physical activity and dietary habits.

OTHER OUTCOMES:
Social Determinants of Health | 5 months
  The investigators recognize that the structural social determinants of health including income inequality, local wealth, sex and ethnic inequalities are key aspects to adolescent health in Aboriginal adolescents. The investigators also recognize that these are unlikely to change with the AYMP. Therefore the investigators will focus on a series of proximal factors. Using Indigenous approaches (i.e. sharing circles, storytelling) the investigators will explore the influence of the AYMP on (1) respect (a major theme in pilot testing), (2) perceived changes in the school environment, (3) family connectedness, (4) peer influence and (5) health behaviours. If youth prefer to discuss issues in a private setting, opportunities will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M McGavock, PhD, Principal Investigator — University of Manitoba, Manitoba Institute of Child Health; Joannie Halas, PhD., Principal Investigator — University of Manitoba
Locations (1):
- Children's Hospital Research Institute of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Eskicioglu P, Halas J, Senechal M, Wood L, McKay E, Villeneuve S, Shen GX, Dean H, McGavock JM. Peer mentoring for type 2 diabetes prevention in first nations children. Pediatrics. 2014 Jun;133(6):e1624-31. doi: 10.1542/peds.2013-2621. Epub 2014 May 12. PMID 24819579